CLINICAL TRIAL: NCT02724982
Title: Body Image Satisfaction In Relation To Body Mass Index And Self- Esteem Among Chinese Female Students: A Cross Sectional Study
Brief Title: Body Image Satisfaction In Relation To Body Mass Index And Self- Esteem Among Chinese Female Students
Status: Completed | Type: Observational
Sponsor: Manisha Parai (Other)
Responsible Party: Sponsor-Investigator, Manisha Parai, Lecturer, Universiti Tunku Abdul Rahman
Organization: Universiti Tunku Abdul Rahman (Other)
Other Study IDs: U/SERC/85/2015
Record Dates: First submitted 2016-01-05; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Self esteem; Body mass index

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
Body image satisfaction and self- esteem level are important to be known among students in order to intervene in a correct time. Body dissatisfaction is one of the factors leading to negative self-perception, low mood, depression, and eating disorders. This may be detrimental to students in their academic performance. However, the correlations of body image satisfaction towards body mass index and self- esteem among university female students are still unclear in Malaysia. Thus, the purpose of this study is to determine its relationships among Chinese female students. university female participants will be included with convenience sampling method. Participants will completed Ronsenberg Self- Esteem Scale and 8 items version of Body Shape Questionnaire. These 2 scales used to measure level of self- esteem and body image satisfaction. Body mass index will be calculated from self- reported height and weight. The data will be analysed by using descriptive and correlation methods.

ELIGIBILITY:
Inclusion Criteria:

* Female and Chinese students
* Age more or equal than 20 years ( ≥20 )
* UTAR students

Exclusion Criteria:

* Male and non-Chinese students
* Age less than 20 ( <20 )
* Non- UTAR students

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chinese female university students in UTAR, Sungai Long campus, Malaysia
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Ronsenberg Self- Esteem Scale | Baseline
body image satisfaction questionnaire | Baseline
Body mass index | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia